CLINICAL TRIAL: NCT01960309
Title: Minimal Invasive Imaging of Coronary Artery Disease in Patients With Asymptomatic Myocardial Injury After Major Non-cardiac Surgery.
Acronym: AMI-NCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Wilton A van Klei, W.A. van Klei, MD PhD, UMC Utrecht
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AMI-NCS
Record Dates: First submitted 2013-07-30; First posted 2013-10-10 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Myocardium; Injury; Coronary Artery Disease
MeSH Terms: conditions — Wounds and Injuries; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1. TnI elevation (Experimental): TnI 0.06-0.60ng/ml, no ischemia on ECG. Intervention: minimal invasive cardiac imaging
  Interventions: Other: Minimal invasive cardiac imaging
- 2. TnI elevation (Experimental): TnI 0.61-6.00 ng/ml, no ischemia on ECG. Intervention: minimal invasive cardiac imaging
  Interventions: Other: Minimal invasive cardiac imaging
- 3. TnI elevation (Experimental): TnI>6.00 ng/ml, no ischemia on ECG. Intervention: minimal invasive cardiac imaging
  Interventions: Other: Minimal invasive cardiac imaging
- 4. TnI elevation (Experimental): TnI >6.00 ng/ml, ischemia on ECG and Hb<5.1. Intervention: minimal invasive cardiac imaging
  Interventions: Other: Minimal invasive cardiac imaging
- 5. TnI elevation (Experimental): TnI >6.00 ng/ml, ischemia on ECG and Hb>5.0. Intervention: minimal invasive cardiac imaging
  Interventions: Other: Minimal invasive cardiac imaging
- Control (Active Comparator): TnI <0.06 ng/ml, no ischemia on ECG. Intervention: minimal invasive cardiac imaging
  Interventions: Other: Minimal invasive cardiac imaging

INTERVENTIONS:
Other: Minimal invasive cardiac imaging — * Coronary CT angiography (CCTA)
  * Coronary magnetic resonance imaging (CMR)
  * Echocardiography

SUMMARY:
This is a cross-sectional pilot study to assess coronary artery disease with minimal invasive techniques in patients with asymptomatic troponin elevation after noncardiac surgery. The primary objective is to quantify coronary artery disease, as determined by coronary CT and MR, as a cause of postoperative myocardial injury. The secondary objective is to correlate coronary calciumscore to postoperative levels of troponin.

ELIGIBILITY:
Inclusion Criteria:

* Major noncardiac surgery with a planned minimal postoperative hospital stay of 2 days
* Age > 59 years
* Troponin_I elevation > 0.06 ng/ml in the first 3 post-operative days
* No clinical symptoms of myocardial ischemia

Exclusion Criteria:

* Perioperative troponin elevation due to other factors than coronary artery disease such as proven pulmonary embolism or sepsis
* Perioperative ST-elevation myocardial infarction (STEMI)
* Perioperative symptomatic angina with troponin elevation
* Patients with a history or ECG-signs of myocardial infarction
* Patients with pre-existent heart failure, left ventricular dysfunction, significant valvular disease or left ventricle hypertrophy
* Patients with significant valvular disease or left ventricle hypertrophy determined postoperatively with echocardiography.
* Contra-indication for CMR such as claustrophobia or metal prosthesis
* Allergic reaction to CT-contrast or gadolinium
* Renal dysfunction with GFR < 50 ml/min, as determined after the operation
* Unstable hemodynamics or other conditions disabling transport to the Radiology department
* Expected major discomfort or substantial increase in pain sensation by undergoing CCTA or CMR
* Admission at the ICU
* Poor prognosis due to other medical conditions e.g. malignancy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-06 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Coronary artery disease | During hospital admission
  Coronary artery disease with luminal narrowing > 50 % in one or more major epicardial vessels by CCTA.

SECONDARY OUTCOMES:
Coronary calcium score | During hospital admission
  Agatston coronary calcium score
Extent of coronary artery atherosclerosis | During hospital admission
  Presence and extent of coronary artery atherosclerosis as measured with coronary CCTA
Minimal myocardial injury | During hospital admission
  Minimal myocardial injury measured by late gadolinium enhancement on CMR.

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik M. Nathoe, MD PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands